CLINICAL TRIAL: NCT02641743
Title: Increased Insulinogenic Indexes Following Liquid Food (Inslow) Intake in Impaired Glucose Tolerance and Type-2 Diabetic Subjects.
Brief Title: Clinical Trial for Liquid Food (Inslow)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Meiji Health Science and Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0001
Record Dates: First submitted 2015-12-20; First posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inslow (Experimental): Each participant was requested to consume one of is energetic test meals (200 kcal per serving 200ml) Inslow at 7:00 AM.
  Interventions: Dietary Supplement: Inslow
- standard balanced formula (Placebo Comparator): Each participant was requested to consume one of is energetic test meals (200 kcal per serving 200ml) standard balanced formula at 7:00 AM.
  Interventions: Dietary Supplement: standard balanced formula

INTERVENTIONS:
Dietary Supplement: Inslow — carbohydrate adjusted liquid food using palatinose as the major carbohydrate (>50%)
  Arms: Inslow
Dietary Supplement: standard balanced formula
  Arms: standard balanced formula

SUMMARY:
A carbohydrate adjusted liquid formula (Inslow) using palatinose as the major carbohydrate (>50%) was devised. Consumption Inslow for a long term (3-5 months) is reported to improve glycemic control by reducing the postprandial plasma glucose levels in diabetes and impaired glucose-tolerant subjects (IGT). The present study intends to understand the mechanism on postprandial glycemic responses.

DETAILED DESCRIPTION:
The test enteral nutrition formula (Inslow) and the standard balanced formula (Meibalance) were administered in a randomized crossover design to 11 healthy people, 13 IGT and 12 type-2 diabetes, judged by the postprandial state after in taking the two test meals in a random order with a washout period of one week. On the day prior to the test day, subjects were asked to stay at the same facility and to take the same supper with 450 kcal controlled, after 21:00 with only water allowed as ad libitum and not do any exercise. Each participant was taken a fasting blood sample, and then requested to consume one of is energetic test meals (200 kcal per serving) Inslow or standard balanced formula at 7:00 AM. Subsequent blood samples were collected at 30,60,90,and 120 min after meal consumption. The plasma concentrations of glucose, insulin, and free fatty acids were measured for each blood sample. Plasma glucose was measured by hexokinase method, plasma insulin by serum radioimmunoassay method and plasma free fatty acid by enzyme chemical method.Routine blood test and biochemical test were performed using the same blood sample only at fasting stage,including RBC, WBC, TP, ALP, T-Cho, etc., to confirm the status of each subject. Collected blood was applied to analyses at Shanghai Meizhong Clinical Measurement Centre. The enteral nutrition meal Inslow was designed by palatinose, dextrin and fiber as carbohydrate for 56%,23% and 15%, respectively. The standard balanced meal was included dextrin as the main carbohydrate for 85%, together with sugar and fiber.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (symptoms of diabetes plus fasting plasma glucose level higher than 7.0 mmol/L and glucose levels after 75g oral glucose tolerance test (OGTT) or casual blood glucose level higher than 11.1mmol/L) and IGT patients (glucose levels after 75g OGTT between 7.8 and 11.1mmol/L).

Exclusion Criteria:

* These patients or subjects have no infectious diseases and were not using any drug.

Ages: 52 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
plasma glucose concentration | 2 weeks

SECONDARY OUTCOMES:
plasma insulin concentration | 2 weeks
plasma free fatty acid concentration | 2 weeks

IPD SHARING:
Plan to Share IPD: No